CLINICAL TRIAL: NCT05472532
Title: Evaluation of an Automated System to Culture Metastatic Patient Circulating Tumor Cells in Embryonated Chicken Eggs (in Ovo Culture)
Acronym: INOVOLINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0492
Record Dates: First submitted 2022-07-07; First posted 2022-07-25 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cancer Metastatic; Prostate Cancer; Breast Cancer; Lung Cancer; Ovarian Cancer; Gastric Cancer
Keywords: chick embryo chorioallantoic membrane; in ovo technology; cancer; Metastatic cancer; CTC; process automation
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms; Breast Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6 cohort (Experimental): Prostate Cohorte : Castrate resistant metastatic prostate cancer patient Breast cohort : HER2+ ou RH+ metastatic breast cancer patient Lung cohort : Non-small cell lung metastatic lung cancer patient Ovarian cohort : Ovarian cancer with peritoneal carcinomatosis Colorectal cohort : Colorectal cancer with peritoneal carcinomatosis Gastric cancer : Gastric cancer with peritoneal carcinomatosis
  Interventions: Procedure: Patient sampling.

INTERVENTIONS:
Procedure: Patient sampling. — One or several bio-specimens will be sampled depending on the cohort :
  * Blood (40 ml)
  * Pleural Fluid (40 ml)
  * Peritoneal liquid (40 ml)
  * Solid tumors

SUMMARY:
A variety of in vivo experimental models have been established for the studies of human cancer using both cancer cell lines and patient-derived xenografts (PDXs). In order to meet the aspiration of precision medicine, the in vivo murine models have been widely adopted. However, common constraints such as high cost, long duration of experiments, and low engraftment efficiency remained to be resolved. The chick embryo chorioallantoic membrane (CAM) is an alternative model to overcome some of these limitations. The chick CAM is shown to be a robust model for both the inoculation of cell lines and grafting of patient tumors for drug therapy evaluations and target genes/pathways analysis.

The start-up INOVOTION has developed a unique, highly sensitive and reproducible CAM assay to graft human cancer cells/tumors in the chicken egg environment. INOVOTION's technology was validated for over 55 human tumor cell lines, including carcinomas, gliomas and melanomas, as well as over 30 reference drugs currently on the market.

At INOVOTION, the graft of human cancer cells on the chicken CAM is currently conducted manually. To scale-up, the process was recently automated. The automation performance was assessed on cancer cells lines. The objective of this study is to demonstrate that the automation of the INOVOTION process enables tumors' proliferation using patient samples (from tumor samples or circulating tumor cells) as grafting material.

ELIGIBILITY:
* Inclusion Criteria for all cohorts * :

  * Age > 18
  * Signed consent
  * Inclusion criteria for the "Prostate" cohort:
  * prostate adenocarcinoma histologically proven
  * metastatic situation
  * at least 2 metastatic sites
  * Evolutionary disease that requires a new treatment
  * Inclusion criteria for the "Breast" cohort:
  * HER2+ or RH+ breast adenocarcinoma histologically proven
  * metastatic situation
  * at least 2 metastatic sites
  * Evolutionary disease that requires a new treatment
  * Inclusion criteria for the "Lung" cohort:
  * Non Small Lung cancer histologically proven
  * metastatic situation
  * at least 2 metastatic sites
  * Evolutionary disease that requires a new treatment
  * Inclusion criteria for "Ovarian" cohort:
  * Ovarian cancer histologically proven
  * Presence of peritoneal carcinomatosis (stage IIIC or IV); with or without presence of peritoneal fluid
  * Inclusion criteria for "Colo-Rectal" cohort:
  * Colo-rectal cancer histologically proven
  * Presence of peritoneal carcinomatosis, with or without presence of peritoneal fluid
  * Evolutionary disease that requires a new treatment
  * Inclusion criteria for "Gastric" cohort:
  * Gastric cancer histologically proven
  * Presence of peritoneal carcinomatosis, with or without presence of peritoneal fluid
* Exclusion Criteria for all cohorts * :

  * Weight <50kg
  * Parallel participation in a doubled blinded study
  * Brain or ganglionary metastasis only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
The main primary endpoint will be reached, if the xenograft rate using patients' samples is ≥ 50% with the INOVOTION automated process. | The sample outcome will be measured 19 days after egg engraftment.
  A xenograft will be considered successful if proliferating human material is found in at least one of the egg engrafted with the patient sample (one patient sample being able to be used to engraft several eggs).
  Success = at least one successful xenograft on all engrafted eggs with a patient sample Failed: 0 successful xenograft on all engrafted eggs with a patient sample

SECONDARY OUTCOMES:
Measure of the xenograft rate per patient sub-population and per cohort (patient blood CTC, pleural fluid, peritoneal fluid, tumor pieces) | The sample outcome will be measured 19 days after egg engraftment
  A xenograft will be considered successful if proliferating human material is found in at least one of the egg engrafted with the patient sample (one patient sample being able to be used to engraft several eggs).
  Success = at least one successful xenograft on all engrafted eggs with a patient sample Failed: 0 successful xenograft on all engrafted eggs with a patient sample
Biological characteristics of the obtained xenografts (per cohort) | One to two months after egg engrafting
  NGS xenograft analysis
Study of xenograft biological responses under different cancer drug treatment (per cohort) | 19 days after egg engraftment.
  biological responses analysis.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Lyon Sud - Department of Medical Oncology, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No